CLINICAL TRIAL: NCT02881450
Title: Prevalence of Inflammatory Myopathies in Alsace
Brief Title: Epidemiological Study of Inflammatory Myopathies in a French Region
Acronym: PREMIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4963
Record Dates: First submitted 2013-12-19; First posted 2016-08-29 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Polymyositis
MeSH Terms: conditions — Polymyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Knowledge of the descriptive epidemiology of MIs is very limited. The main objective of this study is to determine the prevalence of inflammatory myopathies in Alsace at the 1st January 2012 with "capture-recapture" design using several independent sources of case identification.

DETAILED DESCRIPTION:
Inflammatory myopathies (MIs) are a group of muscle diseases with a significant heterogeneity, clinical, immunological and prognosis.

The old classifications, still currently used, highlight this heterogeneity. Therefore Troyanov and coll. and Hoogendijk and coll. have each recently proposed a classification based on clinical and serological - and immuno- histological examination.

The pathogenesis and prognosis of MIs is very different depending on the entity in question.

Knowledge of the descriptive epidemiology of MIs is very limited. In fact no epidemiological work using criteria consensual classification is actually started.

We propose an epidemiological study of MIs. The main objective of the study is to determine the prevalence of MIs in Alsace at 1stJanuary 2012 by means of a "capture- recapture" study using several independent sources of case identification. The secondary objectives of the study are:

* estimating the geographical distribution of the disease in the Alsace region and / or Auvergne
* demographic description of patients : age, sex, residence , occupation
* description of the disease: patient age at diagnosis, disease classification , main clinical manifestations and complications
* Identification of paraneoplastic forms will be for the Alsace region by crossing with Alsatian cancer registries. These records will be interviewed to identify cases of MIs associated with cancers.

ELIGIBILITY:
Inclusion Criteria:

* All patient reported suffering from inflammatory myopathy
* Meeting the Hoogendijk, Troyanov and Griggs classification criteria
* Alive at 1st January 2012- Domiciled in Alsace (Bas-Rhin or Haut-Rhin counties of France)

Exclusion Criteria:

* All patient reported with a different or incomplete diagnosis of inflammatory myopathy (not meeting the Hoogendijk, Troyanov and Griggs criteria)
* All patient dead and/or non-domiciled in Alsace at 1st January 2012

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Resident of Alsace region located in North-east France
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2012-01; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Estimate the prevalence of idiopathic inflammatory myopathies in Alsace. | Prevalence of idiopathic inflammatory myopathies in Alsace at 1st January 2012

CONTACTS AND LOCATIONS:
Overall Officials: Jean SIBILIA, MD, Principal Investigator — University Hospital, Strasbourg, France